CLINICAL TRIAL: NCT02167724
Title: Multicentre Evaluation of Bucco-dental Health in Patients With Schizophrenia in Côte d'Or
Acronym: BUCCODOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DENIS CHS 2014
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Blood Specimen Collection

ARMS (1):
- Patients with schizophrenia (Experimental)
  Interventions: Other: Bucco-dental examination; Other: Blood sample; Other: Clinical and social questionnaire

INTERVENTIONS:
Other: Bucco-dental examination
Other: Blood sample
Other: Clinical and social questionnaire

SUMMARY:
The aim of this study is to know the bucco-dental status of patients with schizophrenia in Côte d'Or.

Participation in this study will last only as long as it takes to:

* carry out a bucco-dental examination: evaluation of dental plaque and calculus
* take a blood sample to assess needs in vitamin C (only for patients included at DIJON CHU and CHS Chartreuse)
* complete a 30-minute questionnaire: clinical data and answers to questions concerning dental hygiene and eating habits.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided consent
* Patients over 18 years of age
* Persons with schizophrenia according to the ICD 10 criteria and followed in hospital (complete or day hospital) in one of the hospitals taking part in the study

Exclusion Criteria:

* Adult under guardianship
* Patient not covered by national health insurance
* Pregnant or breast-feeding women
* Patients not stabilized from a psychiatric viewpoint
* Patients experiencing an acute psychiatric episode
* Impossibility to understand and /or poor understanding of French

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Calculate the DMF index (Decayed, Missing, Filled) | Baselines

SECONDARY OUTCOMES:
Calculate the simplified Oral Health Index (OHI-S) | Baselines
Perception of oral health of patients observed | Baselines

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHS La Chartreuse, Dijon
  - CHU de DIJON, Dijon
  - CH Semur-en-Auxois, Semur-en-Auxois

REFERENCES:
- [Result] Denis F, Milleret G, Wallenhorst T, Carpentier M, Rude N, Trojak B. Oral health in schizophrenia patients: A French Multicenter Cross-Sectional Study. Presse Med. 2019 Feb;48(2):e89-e99. doi: 10.1016/j.lpm.2018.06.018. Epub 2019 Mar 8. PMID 30853291